CLINICAL TRIAL: NCT02241252
Title: Clinical Validation of an iPhone ECG System, QT Substudy
Brief Title: Using an iPhone ECG to Monitor the QT Interval on Dofetilide and Sotalol Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OU_IRB_3237
Record Dates: First submitted 2014-09-08; First posted 2014-09-16 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Cardiac Arrhythmia; Qt Interval, Variation in
Keywords: ECG; QT interval; Sotalol; Dofetilide; iPhone
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- iPhone ECG QT recording (Other): iPhone ECG
  Interventions: Device: iPhone ECG

INTERVENTIONS:
Device: iPhone ECG — Please see detailed description for additional information.
  Other Names: AliveCor iPhone ECG

SUMMARY:
This study will validate the recording accuracy of a specific electrical interval of the heart, the QT interval, between an iPhone rhythm strip recording and a traditional 12-lead electrocardiogram (ECG). These measurements will occur in hospitalized patients that are starting either sotalol or dofetilide, since both of these medications can prolong the QT interval.

DETAILED DESCRIPTION:
Patients that were already selected to begin either dofetilide or sotalol in the hospital, will be included in the study. Patients will receive an ECG before and 2 hours after each dose of the medication, which is done to monitor the QT interval. In addition, patients that consent to participate in the study will have an iPhone ECG recording taken in lead positions that correspond to leads I,II, and III.

These recordings will be compared and analyzed to assess the accuracy of the QT interval recordings between the two methods.

ELIGIBILITY:
Inclusion Criteria:

* initiation of sotalol or dofetilide
* inpatient at University hospital

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
QT interval measurement (in milliseconds) | Participants will be followed for duration of hospital stay during which dofetilide or sotalol are being started, an expected average of 3 days
  The QT interval (measured from the start of the QRS to the end of the T wave) will be measured on the 12-lead ECG and on the iPhone rhythm strip recording. Both measurements will be recorded in milliseconds and will be statistically analyzed for bias and agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Garabelli, MD, Principal Investigator — University of Oklahoma; Dwight W Reynolds, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States